CLINICAL TRIAL: NCT03146013
Title: Evaluation of the MP Diagnostics HTLV Blot 2.4
Brief Title: Dual Algorithm Post Market Clinical Study
Status: Completed | Type: Observational
Sponsor: MP Biomedicals, LLC (Industry)
Collaborators: MP Biomedicals Asia Pacific Pte. Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: MP EIA-HTLV-001B Amendment 6.0
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: HTLV-I Infections; HTLV-II Infections; Human T-lymphotropic Virus 1; Human T-lymphotropic Virus 2; HTLV I Associated T Cell Leukemia Lymphoma; HTLV I Associated Myelopathies
Keywords: HTLV; Confirmatory; Supplemental; Blot; HTLV-I; HTLV-II
MeSH Terms: conditions — HTLV-I Infections; HTLV-II Infections; Leukemia-Lymphoma, Adult T-Cell; Paraparesis, Tropical Spastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- HTLV Repeat Reactive (RR) / Non Reactive (NR): Blood donor specimens that tested repeat reactive on the first FDA licensed HTLV screening assay and non-reactive on the second FDA licensed HTLV screening assay
  Interventions: Diagnostic Test: MP Diagnostics HTLV Blot 2.4

INTERVENTIONS:
Diagnostic Test: MP Diagnostics HTLV Blot 2.4 — HTLV I/II Confirmation and Differentiation
  Other Names: HTLV I/II Western Blot Assay

SUMMARY:
The purpose of this study is to assess the validity and reproducibility of the MP Diagnostics HTLV Blot 2.4 in blood specimens testing repeat reactive (RR) on the first FDA licensed screening assay (Abbott Prism) and non-reactive (NR) on the second FDA licensed screening assay (Avioq ELISA).

DETAILED DESCRIPTION:
This is a prospective study designed to assess the safety and effectiveness of a dual algorithm testing for HTLV I/II in blood donors. The study hypothesis is that blood donors testing repeat reactive (RR) on the first FDA licensed HTLV screening assay and non-reactive (NR) on a second FDA licensed screening assay will be confirmed as indeterminate or negative on the MP Diagnostics HTLV Blot 2.4.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Completion of a health history evaluation for routine donor screening
3. Provided a routine blood donation
4. Tests repeat reactive by the Abbott PRISM HTLV assay and non-reactive on the AVIOQ Elisa HTLV assay

Exclusion Criteria:

1. Unwilling or unable to provide informed consent to blood donation
2. Inadequate sample volume for testing
3. Unable to provide samples that meet the suitability requirements for testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All populations are from whole blood donors.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Assess the HTLV dual algorithm testing in blood donor facilities | 3 months
  HTLV I/II confirmation of specimens testing RR on the first FDA licensed HTLV screening assay and non-reactive (NR) on a second FDA licensed HTLV screening assay.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stramer, Ph.D, Principal Investigator — American National Red Cross
Locations (1):
- American Red Cross - National Testing Laboratory, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) was deidentified prior to sharing.

REFERENCES:
- [Background] Miller L. Profile of the MP Diagnostics HTLV Blot 2.4 test: a supplemental assay for the confirmation and differentiation of antibodies to HTLV-1 and HTLV-2. Expert Rev Mol Diagn. 2016;16(2):135-45. doi: 10.1586/14737159.2016.1123622. Epub 2016 Jan 11. PMID 26589659